CLINICAL TRIAL: NCT05300256
Title: Peripheral Heating and Glucose Tolerance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Jeffrey Moore, Adjunct Professor, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PHTGLUCOSE
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Glucose Tolerance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peripheral Heating (Experimental): Peripheral Heating
  Interventions: Device: Peripheral Heating
- Sham (Sham Comparator): Sham
  Interventions: Device: Sham

INTERVENTIONS:
Device: Peripheral Heating — Peripheral heating of the feet
  Arms: Peripheral Heating
Device: Sham — Sham
  Arms: Sham

SUMMARY:
Effect of peripheral heating on glucose tolerance

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years

Exclusion Criteria:

* Open wounds on feet or legs
* Peripheral neuropathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Glucose concentrations | 1 hour

SECONDARY OUTCOMES:
Insulin concentrations | 1 hour
Blood flow | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States